CLINICAL TRIAL: NCT01149083
Title: Phase II Trial of Single Agent ABT-888 With Post-Progression Therapy of ABT-888 in Combination With Carboplatin in Patients With Stage IV BRCA-Associated Breast Cancer
Brief Title: Veliparib With or Without Carboplatin in Treating Patients With Stage III or IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01379; NCI-2011-01379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-96; CHNMC-PHII-96; CDR0000674384; 8264 (Other: City of Hope Comprehensive Cancer Center); 8264 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00039 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); N01CM62201 (NIH); N01CM62202 (NIH); N01CM62203 (NIH); N01CM62209 (NIH); P30CA033572 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Unresectable Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Specimen Handling; Carboplatin; Magnetic Resonance Spectroscopy; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase II (veliparib, carboplatin) (Experimental): Patients receive veliparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Upon progression, patients are taken off treatment for 1 week and may then continue to recieve veliparib along with carboplatin IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Veliparib
- Safety Lead-In Phase (veliparib, carboplatin) (Experimental): Patients receive veliparib PO BID twice daily on days 1-21 of each cycle and carboplatin IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Veliparib

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase II trial studies how well veliparib with or without carboplatin works in treating patients with stage III or IV breast cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether veliparib is more effective with or without carboplatin in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of single agent veliparib (ABT-888) (NSC 737664) in breast cancer (BRCA) carriers with metastatic breast cancer based on response rate (Response Evaluation Criteria In Solid Tumors [RECIST] criteria).

SECONDARY OBJECTIVES:

I. To conduct subset analysis on BRCA1 versus (vs.) BRCA2 and hormone receptor status.

II. To evaluate progression-free survival of patients on single-agent ABT-888. III. To further describe the safety and tolerability of ABT-888 (NSC 737664) as a single agent and in combination with carboplatin for BRCA-associated breast cancer.

IV. To evaluate the pharmacokinetics of ABT-888 (NSC 737664) alone and in combination with carboplatin.

V. To assess the relationship between the level of poly adenosine diphosphate (ADP) ribose polymerase (PARP) inhibition by ABT-888 and biomarkers of deoxyribonucleic acid (DNA) damage in peripheral blood mononuclear cell (PBMC's) and in tumor.

VI. To explore the relationship between biomarkers of drug effect and progression-free survival.

VII. To evaluate the efficacy and safety of the combination of carboplatin and ABT-888 in patients who have failed single agent ABT-888.

VIII. To conduct subset analysis on BRCA1 vs. BRCA2 and hormone receptor status.

OUTLINE: This is a dose-escalation study of veliparib. Patients are assigned to 1 of 2 phases.

SAFETY LEAD-IN PHASE: Patients receive veliparib orally (PO) twice daily (BID) on days 1-21 of each cycle and carboplatin intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.

PHASE II: Patients receive veliparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Upon progression, patients are taken off treatment for 1 week and may then continue to recieve veliparib along with carboplatin IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.

* As of the November 9, 2023 amendment, the pharmaceutical collaborator has discontinued the ABT-888 development program with the National Cancer Institute Cancer Therapy Evaluation Program (CTEP). Clinical supply will no longer be available after December 31, 2024. Patients will discontinue treatment by December 31, 2024, or earlier.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female, and must have histologically confirmed breast cancer that is metastatic or locally advanced, unresectable and for which standard curative measures do not exist or are no longer effective
* Patients must have a known deleterious BRCA mutation confirmed by report from a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory (generally Myriad Genetics Laboratory). It is expected that BRCA testing will be covered as medically necessary care by the patient's insurance carrier
* Measurable disease by RECIST criteria; (evaluable disease is allowed only for the safety lead-in phase)
* Prior chemotherapy regimens for metastatic disease are completed, at least 3 weeks prior to starting therapy; prior radiation and hormonal treatment must be completed at least 1 week prior to starting therapy
* Female, age >= 18 years. Because no dosing or adverse event data are currently available on the use of ABT-888 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of greater than four months
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 times institutional upper limit of normal
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 times institutional upper limit of normal unless there is evidence of liver metastasis, in which case the AST (SGOT)/ALT (SGPT) must be =< 5 times institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* If a woman is of child-bearing potential, a negative serum or urine pregnancy test is required; (The effects of ABT-888 [NSC 737664] on the developing human fetus are unknown; for this reason and because PARP Inhibitor agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; participants should agree to use contraception for at least 3 months after the completion of study therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior therapy with platinum agents (adjuvant therapy with platinum agents is allowed, if completed >= 12 months prior to relapse), or PARP inhibitors (prior iniparib, since it is no longer considered a PARP inhibitor, is allowed)
* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) metastases requiring anticonvulsive medications, or steroids or with active symptomatology; patients on anticonvulsant medications prescribed for reasons other than CNS metastases, not on steroids and without active symptomatology are eligible; patients must be off anti-seizure medications and steroids for 3 months or more before enrollment
* Patients with active seizure or a history of seizure; patients with CNS metastases must be stable after therapy for > 3 months and off steroid treatment prior to study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biological composition to ABT-888 (NSC 737664) or PARP inhibitors
* Patients with contraindications to platinum agents are excluded
* Prior or current non-breast malignancy within 5 years except non-melanoma skin cancer or resected stage I ovarian cancer
* Patients with any non-malignant intercurrent illness (e.g., cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment or which is of such severity that the investigators deem it unwise to enter the patient on protocol
* Pregnant women are excluded from this study because ABT-888 (NSC 737664) has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ABT-888 (NSC 737664), breastfeeding should be discontinued
* Patients unable to swallow the ABT-888 tablets whole are ineligible; (the tablets cannot be crushed or broken)
* Patients with an active severe infection; known infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus; HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ABT-888 (NSC 737664); in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (23):
- United States (22):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Egger SJ, Chan MMK, Luo Q, Wilcken N. Platinum-containing regimens for triple-negative metastatic breast cancer. Cochrane Database Syst Rev. 2020 Oct 21;10(10):CD013750. doi: 10.1002/14651858.CD013750. PMID 33084020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 patients were enrolled in the Phase I trial and 49 patients in the Phase II trial. However, 5 were either inevaluable or did not start treatment, resulting in 44 patients included in the final sample. Of those 5 patients, 3 did not get any drug due to consent withdrawal or choosing other therapy. The remaining 2 were treated but were deemed inevaluable due to not receiving enough drug per protocol. Hence there is data sent to the NCI on those 2 patients who were not part of the analysis.
Groups:
- Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I): Patients receive veliparib 50 mg PO BID on days 1-21 of each cycle and carboplatin AUC 6 IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
- Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I): Patients receive veliparib 50 mg PO BID on days 1-21 of each cycle and carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
- Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I): Patients receive veliparib 100 mg PO BID on days 1-21 of each cycle and carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
- Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I); Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II); Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II): Patients receive veliparib 150 mg PO BID on days 1-21 of each cycle and carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
- Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I): Patients receive veliparib 200 mg PO BID on days 1-21 of each cycle and carboplatin AUC 5 IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
Period: Overall Study
Arm/Group | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II)
Started | 7 | 6 | 3 | 6 | 6 | 24 | 22
Completed | 7 | 6 | 3 | 6 | 6 | 22 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II) | Total
Number analyzed (Participants) | 7 | 6 | 3 | 6 | 6 | 22 | 22 | 72
Age, Continuous [Median (Full Range); unit: Years] | 47 [41 to 62] | 53 [41 to 65] | 44 [34 to 44] | 52 [33 to 66] | 44 [32 to 64] | 42 [28 to 68] | 44 [28 to 67] | 43 [28 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 6 | 6 | 22 | 22 | 72
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Black | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 8
  Caucasian | 6 | 6 | 2 | 5 | 6 | 11 | 5 | 41
  Hispanic | 1 | 0 | 1 | 1 | 0 | 4 | 15 | 22
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 3 | 6 | 6 | 22 | 22 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm; Partial Response (PR), at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; Overall Response (OR) = CR + PR
Time Frame: Up to 8 weeks post-treatment
Population: Arm A includes all patients across dose levels (DL1-DL5) in the safety lead-in Phase I portion of the study, while Arm B comprises only BRCA1 and BRCA2 mutation carriers in the Phase II portion. The protocol pre-specified that the response rate for Phase I would be collected and reported as a single arm/group.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A - Safety Lead-in (Phase I): Patients receive a starting dose of 50 mg veliparib PO BID on days 1-21 of each cycle and 5 AUC carboplatin IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
Arm/Group | Arm A - Safety Lead-in (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II)
Number analyzed (Participants) | 27 | 22 | 22
Participants | 15 | 3 | 8

2. Primary Outcome: Progression-free Survival
Description: Progression-free survival will be summarized as time from first protocol treatment until progression or death from any cause, using the product-limit Kaplan-Meier estimator. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From start of treatment to time of progression or death from any cause, whichever occurs first, assessed up to at least 1 year
Population: Arm A includes all patients across dose levels (DL1-DL5) in the safety lead-in Phase I portion of the study, while Arm B comprises only BRCA1 and BRCA2 mutation carriers in the Phase II portion. The protocol pre-specified that progression-free survival for Phase I would be summarized and reported as a single arm/group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Safety Lead-In (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II)
Number analyzed (Participants) | 27 | 22 | 22
Months | 8.7 [7.3 to 10.6] | 3.6 [2.0 to 6.4] | 6.6 [5.2 to 9.6]

3. Secondary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose of veliparib in combination with AUC 5 of Carboplatin is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 21 days from start of treatment, up to 2 years
Measure: Number; unit: mg
Groups:
- Safety Lead-In (Phase I): Patients receive a starting dose of 50 mg veliparib PO BID on days 1-21 of each cycle and 5 AUC carboplatin IV over 30 minutes on day 1 of each cycle. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and may optionally undergo biopsies throughout the study. Patients undergo blood sample collection during screening and on study.
Arm/Group | Safety Lead-In (Phase I)
Number analyzed (Participants) | 28
mg | 150

4. Secondary Outcome: Number of Participants With at Least One Dose Limiting Toxicity (DLT) - Phase I
Description: Dose-limiting toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Pre-specified DLT criteria included the following adverse events (AE), judged to be at least possibly related to study therapy: any grade III non-hematological toxicity not reversible to grade II or less within 96 hours, or any grade IV toxicity (excluding alopecia or controllable nausea and vomiting). Additionally, patients unable to take 80% of the planned ABT-888 due to toxicity/tolerability will be considered to have had a DLT.
Time Frame: During the first cycle of treatment, up to 21 days
Population: This is a Phase I/II trial with the Phase I portion designed to determine the maximum tolerated dose of veliparib in combination with carboplatin. Arm A is separated into 5 different dose levels to adequately evaluate DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I)
Number analyzed (Participants) | 7 | 6 | 3 | 6 | 6
Participants | 2 | 1 | 0 | 0 | 3

5. Secondary Outcome: Overall Survival
Description: Overall survival will be summarized as time from first protocol treatment until death from any cause, using the product-limit Kaplan-Meier estimator.
Time Frame: From start of treatment to time of death from any cause, assessed up to at least 3 years
Population: Arm A includes all patients across dose levels (DL1-DL5) in the safety lead-in Phase I portion of the study, while Arm B comprises only BRCA1 and BRCA2 mutation carriers in the Phase II portion. The protocol pre-specified that outcomes for Phase I would be summarized and reported as a single arm/group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Safety Lead-In (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II)
Number analyzed (Participants) | 27 | 22 | 22
Months | 18.8 [15.0 to 23.2] | 11.9 [11.2 to NA] — The upper confidence limit for overall survival is "not reached". | 14.7 [12 to NA] — The upper confidence limit for overall survival is "not reached".

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 5 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II)
All-Cause Mortality (participants affected / at risk) | 6/7 | 6/6 | 2/3 | 4/6 | 4/6 | 11/22 | 12/22
Serious Adverse Events (participants affected / at risk) | 6/7 | 3/6 | 2/3 | 3/6 | 2/6 | 8/22 | 6/22
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 3/3 | 6/6 | 6/6 | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) (N=7) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=3) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) (N=22) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II) (N=22)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 1 (3) | 1 (2) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A, Dose Level 1 - 50 mg Veliparib, AUC 6 Carboplatin (Phase I) (N=7) | Arm A, Dose Level -1 - 50 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm A, Dose Level A - 100 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=3) | Arm A, Dose Level B - 150 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm A, Dose Level C - 200 mg Veliparib, AUC 5 Carboplatin (Phase I) (N=6) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA I Carriers (Phase II) (N=22) | Arm B - 150 mg Veliparib, AUC 5 Carboplatin BRCA II Carriers (Phase II) (N=22)
Acute kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Allergic reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (85) | 6 (93) | 3 (28) | 6 (137) | 5 (52) | 14 (71) | 18 (111)
Arthralgia (General disorders) | 0 (0) | 1 (1) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 5 (14)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (21)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (8)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 3 (14)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (27) | 0 (0) | 1 (3) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (10)
Dry eye (Eye disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (General disorders) | 2 (4) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 2 (18) | 2 (7)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema cerebral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 1 (2)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (2)
Flank pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Flu like symptoms (General disorders) | 1 (1) | 1 (3) | 1 (1) | 1 (5) | 0 (0) | 1 (1) | 1 (2)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (22)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 3 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6)
Generalized muscle weakness (General disorders) | 3 (3) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 1 (5)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (General disorders) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Investigations) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hyperglycemia (Investigations) | 1 (1) | 4 (20) | 2 (2) | 3 (19) | 2 (2) | 7 (44) | 8 (63)
Hyperhidrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (30) | 0 (0) | 1 (2) | 3 (32)
Hyperkalemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (12) | 2 (3)
Hypermagnesemia (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (4)
Hyperphosphatemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (28) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (22) | 0 (0) | 0 (0) | 1 (3)
Hypoalbuminemia (Investigations) | 2 (2) | 3 (9) | 1 (5) | 3 (9) | 1 (1) | 5 (11) | 5 (21)
Hypocalcemia (Investigations) | 2 (9) | 5 (12) | 2 (22) | 4 (9) | 1 (1) | 6 (20) | 5 (14)
Hypoglycemia (Investigations) | 3 (11) | 2 (4) | 2 (4) | 0 (0) | 1 (1) | 2 (3) | 3 (5)
Hypokalemia (Investigations) | 3 (19) | 2 (7) | 1 (4) | 1 (3) | 0 (0) | 3 (11) | 4 (7)
Hypomagnesemia (Investigations) | 1 (8) | 2 (4) | 1 (2) | 1 (26) | 0 (0) | 0 (0) | 2 (3)
Hyponatremia (Investigations) | 3 (5) | 5 (35) | 2 (5) | 1 (1) | 1 (7) | 4 (9) | 6 (11)
Hypophosphatemia (Investigations) | 1 (4) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 2 (9) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (6) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 2 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 5 (5) | 5 (5)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 5 (8)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Vascular disorders) | 0 (0) | 1 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 5 (12) | 4 (16) | 1 (1) | 1 (37) | 0 (0) | 2 (7) | 4 (31)
Periorbital edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Postnasal drip (General disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Restlessness (General disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shingles (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (8)
Somnolence (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 2 (3) | 2 (6)
Spasticity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombotic thrombocytopenic purpura (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 5 (79) | 5 (99) | 3 (17) | 5 (104) | 5 (49) | 10 (62) | 15 (118)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 3 (7) | 3 (6) | 1 (10) | 0 (0) | 0 (0) | 2 (9) | 5 (21)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 6 (32) | 9 (21)
Constipation (Gastrointestinal disorders) | 6 (23) | 5 (11) | 3 (17) | 4 (8) | 2 (5) | 8 (40) | 14 (59)
Diarrhea (Gastrointestinal disorders) | 4 (7) | 1 (2) | 0 (0) | 1 (11) | 0 (0) | 8 (15) | 10 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (13) | 3 (18)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 3 (10) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (17)
Nausea (Gastrointestinal disorders) | 7 (31) | 6 (25) | 2 (7) | 5 (16) | 5 (22) | 18 (91) | 22 (154)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (13) | 4 (16) | 2 (11) | 3 (7) | 3 (9) | 10 (22) | 17 (62)
Chills (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 4 (4)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (59) | 6 (59) | 3 (17) | 5 (35) | 6 (23) | 14 (98) | 18 (146)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 2 (5) | 5 (7)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pain (General disorders) | 5 (12) | 4 (9) | 2 (5) | 3 (7) | 2 (2) | 4 (33) | 8 (88)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 1 (6) | 1 (1) | 1 (1) | 2 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (17)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Intraoperative head and neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (8) | 2 (20) | 2 (11) | 1 (4) | 8 (28) | 8 (32)
Alkaline phosphatase increased (Investigations) | 3 (5) | 5 (30) | 2 (16) | 3 (56) | 1 (2) | 10 (55) | 11 (41)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 3 (24) | 2 (14) | 3 (15) | 2 (2) | 10 (30) | 11 (32)
Creatinine increased (Investigations) | 0 (0) | 3 (5) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (5)
INR increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (73) | 5 (90) | 3 (16) | 3 (13) | 2 (39) | 9 (54) | 7 (51)
Neutrophil count decreased (Investigations) | 5 (41) | 6 (52) | 3 (5) | 5 (70) | 4 (25) | 10 (44) | 10 (41)
Platelet count decreased (Investigations) | 5 (66) | 6 (83) | 3 (44) | 6 (85) | 6 (48) | 14 (42) | 14 (55)
Weight gain (Investigations) | 1 (9) | 3 (11) | 1 (16) | 1 (16) | 0 (0) | 3 (39) | 5 (25)
Weight loss (Investigations) | 0 (0) | 2 (3) | 0 (0) | 3 (52) | 1 (2) | 2 (3) | 2 (13)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 1 (3) | 2 (3) | 2 (3) | 1 (1) | 5 (17) | 8 (25)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (30) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (10) | 7 (18)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (13) | 2 (5) | 1 (3) | 0 (0) | 2 (2) | 4 (13)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 3 (11) | 0 (0) | 1 (4) | 3 (15)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (3) | 1 (2) | 1 (1) | 3 (20) | 5 (43)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 4 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 2 (5) | 0 (0) | 1 (5) | 3 (5)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (8)
Dizziness (Nervous system disorders) | 2 (7) | 2 (5) | 1 (2) | 2 (8) | 0 (0) | 9 (20) | 13 (31)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (12) | 5 (17) | 3 (6) | 1 (1) | 1 (5) | 7 (22) | 9 (45)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 1 (2) | 1 (8) | 3 (11) | 1 (6) | 3 (8) | 4 (32)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (6)
Agitation (Psychiatric disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (5) | 2 (6) | 2 (3) | 3 (16) | 0 (0) | 4 (8) | 7 (36)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (8) | 0 (0) | 1 (2) | 2 (3) | 1 (2) | 3 (16) | 4 (30)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (3) | 1 (2) | 2 (24) | 0 (0) | 7 (24) | 5 (15)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 2 (4)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (12)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (15) | 2 (18)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2) | 3 (11) | 3 (6) | 0 (0) | 8 (31) | 10 (44)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (9) | 4 (8) | 2 (17) | 1 (3) | 1 (1) | 5 (14) | 8 (37)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (6) | 2 (4) | 3 (29) | 7 (77)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (3) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (6) | 2 (14)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Flushing (Vascular disorders) | 2 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 2 (10) | 2 (6) | 1 (2) | 3 (32) | 1 (1) | 5 (23) | 8 (51)
Hypertension (Vascular disorders) | 1 (12) | 1 (2) | 1 (13) | 2 (70) | 1 (5) | 5 (40) | 4 (24)
Hypotension (Vascular disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT01149083/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT01149083/ICF_001.pdf